CLINICAL TRIAL: NCT00382278
Title: Phase 1/2 Study of Autologous Bone Marrow Derived Mononuclear Cells in Liver Cirrhosis
Brief Title: Safety Study of Autologous Stem Cell in Liver Cirrhosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other authors showed the same metabolic effect may be obtained when BMMC are delivered peripherally, with lower risk and cost than through hepatic artery.
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Guilherme Ferreira da Motta Rezende, UFRJ
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CELTHEP-01
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-02

CONDITIONS: Liver Cirrhosis
Keywords: Stem cell; Liver cirrhosis; Cellular therapy; Autologous; Bone marrow
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Autologous bone marrow-derived mononuclear cells infusion — Under local anesthesia, 100 mL of bone marrow were aspirated from the posterior iliac crest. ABMMC were isolated by density gradient centrifugation in Ficoll-Hypaque gradient, 10% of the cells were labeled with SnCl2-99mTc, and a small fraction was used for cell counting and viability analysis. At least 100 millions of mononuclear-enriched BMC suspended in 20 mL of saline were delivered preferentially in the common hepatic artery by celiac trunk catheterism.

SUMMARY:
It is a fase I/II clinical study to evaluate feasibility, safety and kinetics of cellular therapy with bone marrow-derived mononuclear cells (ABMMC) in patients with liver cirrhosis. All the patients have moderate liver disfunction and a waiting time expectancy of liver transplantation longer than 12 months due their low MELD score. The ABMMC are labeled with 99mTc and infused through the hepatic artery. Scintigraphy is performed 2 and 24 hours after infusion. Patients are submitted to frequent clinical, laboratorial and image evaluation during the follow up period of 12 months.

DETAILED DESCRIPTION:
A one year clinical trial was conducted. Patients had moderate liver dysfunction and a liver transplant was not expected to occur earlier than 12 months, due to low MELD scores. Hepatocellular carcinoma (HCC) and hepatic artery or portal vein thrombosis were excluded by color Doppler ultrasonography (DUS) and 3-phase computed tomography (CT). Under local anesthesia, 100 mL of bone marrow were aspirated from the posterior iliac crest. ABMMC were isolated by density gradient centrifugation in Ficoll-Hypaque gradient, 10% of the cells were labeled with SnCl2-99mTc, and a small fraction was used for cell counting and viability analysis. ABMMC were delivered preferentially in the common hepatic artery by celiac trunk catheterism. Total body scintigraphy (TBS) was performed 3 hours after infusion. Patients were submitted to frequent clinical, biochemical and imaging evaluation during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any origin
* Moderate liver disfunction (Child-Pugh Score=7-10)

Exclusion Criteria:

* Waiting time expectancy of liver transplant shorter than 12 months
* Ongoing hepatic encephalopathy
* Clinically detectable ascitis
* Severe coagulation disorder (INR>2,0 or platelets count < 40.000)
* Diagnosis or strong suspicion of cancer (except basocellular)
* Pregnancy or intention to become pregnant during the next 12 months
* Moderate or severe co-morbidity
* Current participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Changes in liver function according to Child-Pugh and MELD scores | in days 1,2,7,14,30, 45, 60, 90, 120, 150, 180, 270, 360
Hepatic artery and portal vein thrombosis (doppler ultrasound) | in days 1,2,7,14,90, 180 and 360
Development of liver nodule (ultrasound screening) | in days 1,2,7,14,90, 180 and 360 (US) and in day 360 (CT scan )
Liver related mortality | 360 days

SECONDARY OUTCOMES:
Body distribution of 99mTc labeled BMDMC (scintigraphy) | after 3 hours of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme FM Rezende, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil